CLINICAL TRIAL: NCT06099600
Title: Randomized Study Evaluating the Value of a Pre-habilitation Stay and Digital Follow-up, Compared With Standard Management, in Anterior Cruciate Ligament Reconstruction
Brief Title: Anterior Cruciate Ligament Reconstruction
Acronym: Préhab-LCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A01633-42
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Ligament Rupture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-habilitation stays (Experimental): Pre-habilitation involves taking part in a half-day information session led by a physiotherapist and a nurse prior to surgery. Patients will benefit from digital monitoring via the Orthense application, as well as scheduled surgery (anterior cruciate ligament reconstruction) and the usual peri-operative medical follow-up.
  Interventions: Procedure: Reconstructive surgery of the anterior cruciate ligament
- conventional care (Active Comparator): During their pre-operative visit with the surgeon, patients will receive a booklet containing information on the peri-operative period, possible complications, how to prevent them and what to do should they occur. Patients will benefit from standard computerized follow-up, as well as the scheduled surgical procedure (anterior cruciate ligament reconstruction) and the usual peri-operative medical follow-up.
  Interventions: Procedure: Reconstructive surgery of the anterior cruciate ligament

INTERVENTIONS:
Procedure: Reconstructive surgery of the anterior cruciate ligament — surgical reconstruction after rupture of the anterior cruciate ligament is widely proposed as first-line treatment, with the aim of restoring knee joint stability and facilitating functional recovery

SUMMARY:
This study evaluates the effectiveness of a pre-habilitation stay via digital monitoring on patients' short-term post-operative anxiety, compared with conventional management.

DETAILED DESCRIPTION:
This is a prospective, comparative, randomized (2-arm), controlled, single-center study of two management modalities.

Recruitment will focus on adult patients with anterior cruciate ligament rupture and scheduled anterior cruciate ligament surgical reconstruction. Patients will be randomized into 2 arms, an experimental arm A (pre-habilitation management) and a control arm B (conventional management).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ;
* Partial or complete primary anterior cruciate ligament rupture;
* Partial or complete primary rupture of the anterior cruciate ligament;
* Scheduled anterior cruciate ligament reconstructive surgery;
* Patient with a tablet, computer or smartphone with an internet connection;
* Patient able to understand and read French;
* Willingness to complete questionnaires at regular intervals;
* Membership of a social security scheme;
* Signed informed consent.

Exclusion Criteria:

* Recurrence / contralateral lesion ;
* Stage III collateral ligament injury;-
* Osteotomy ;
* Neurological (motor and/or sensory), vestibular or rheumatic pathology;
* Pregnant or breast-feeding woman;
* Protected adult patient (under guardianship, curatorship or deprivation of liberty).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory questionnaire | 7 days
  The main evaluation criterion is the total "state-anxiety" score of the State-Trait Anxiety Inventory questionnaire on 7 days compared to the score measured at least 25 days (i.e. baseline value: before the surgical intervention and before the pre-habilitation stay taking place for patients in the experimental group)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France